CLINICAL TRIAL: NCT00219843
Title: A Phase 1 Safety and Tolerability Study of Intralesional PV-10 Chemoablation in Subjects With Metastatic Melanoma
Brief Title: Intralesional PV-10 Chemoablation of Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PV-10-MM-01
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Melanoma
Keywords: Stage III and IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Rose Bengal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PV-10 (rose bengal disodium, 10%)

SUMMARY:
The objective of this study is to investigate the safety of intralesional (IL) PV-10 for the treatment of metastatic melanoma. This study will also include a preliminary assessment of response of treated and untreated lesions by clinical evaluation at follow-up of 12 to 24 weeks following IL PV-10 treatment.

DETAILED DESCRIPTION:
This is a two center, open label, ascending dose study. Subjects with at least two measurable melanoma lesions will receive a single intralesional injection of 10% PV-10 solution into each of one to twenty (20) target lesions. Additionally, one to three measurable untreated non-target lesions will be followed for assessment of bystander response. Systemic and locoregional adverse events will be monitored over the study interval. Dose escalation will be made only if no subjects at the first dose level have a Grade 3 non-hematological or Grade 4 hematological toxicity over a period of two weeks after PV-10 administration. Subject accrual and PV-10 administration at the second dose level will be stopped if more than 1 subject has a treatment related Grade 3 non-hematological or Grade 4 hematological toxicity within a period of two weeks after PV-10 administration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic melanoma, American Joint Committee on Cancer (AJCC) Stage III (regional lymph node metastasis, in-transit metastasis or satellite metastasis) or Stage IV (distant metastasis)
* Measurable disease in at least two lesions, each lesion ≤ 6 cm in diameter
* Performance status: ECOG 0-2
* Life expectancy: at least 6 months
* Hematopoietic:

  * White blood cell count (WBC) at least 3000/mm3
  * Absolute neutrophil count (ANC) at least 1.5 (1,500/mm3)
  * Platelet count at least 100,000/mm3
* Renal function:

  * Creatinine ≤ 2.0 mg/dL
* Hepatic function:

  * Bilirubin ≤ 2.0 mg/dL
  * AST/ALT ≤ 3 times the upper limit of normal (ULN)
* Cardiovascular function:

  * No major cardiovascular disease
* Thyroid function:

  * T3 (serum triiodothyronine), T4 (serum thyroxine) and THS (serum thyrotropin) within normal limits
* Immunological function:

  * Adequate immune system function in the opinion of the investigator

Exclusion Criteria:

* Radiation therapy within 4 weeks or to any study lesion within 12 weeks
* Chemotherapy or other systemic cancer therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin) or regional chemotherapy (limb infusion or perfusion) within 12 weeks
* Local treatment (e.g., surgery, cryotherapy, radiofrequency ablation) to the treatment area within 4 weeks
* Investigational agents within 4 weeks (or 5 half-lives)
* Anti-tumor vaccine therapy within 12 weeks
* Concurrent illness:

  * Severe diabetes or extremity complications due to diabetes
  * Significant concurrent disease or illness, psychiatric disorders, or alcohol or chemical dependence that would, in the opinion of the investigator, compromise subject safety or compliance or interfere with interpretation of study results
  * Thyroid autoregulatory dysfunction, including thyroid disease (subclinical or ongoing), goiter, partial thyroidectomy, prior radioiodine- or surgically-treated Graves' hyperthyroidism, or cystic fibrosis
  * Pregnancy or fertile female subjects who are not using effective contraception
* Concurrent medications:

  * Subjects taking medications with a significant risk of photosensitization, such as thiazides, within one week (or 5 half-lives) of study treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety: adverse experience

SECONDARY OUTCOMES:
Efficacy: objective response rate of target lesions and untreated non-target lesions

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Pharmaceuticals
Locations (2):
- Australia (2):
  - Sydney Melanoma Unit, North Sydney, New South Wales
  - Newcastle Melanoma Unit, Waratah, New South Wales